CLINICAL TRIAL: NCT02178722
Title: A Phase 1/2 Study Exploring the Safety, Tolerability, and Efficacy of MK-3475 in Combination With INCB024360 in Subjects With Selected Cancers (ECHO-202/KEYNOTE-037)
Brief Title: Study to Explore the Safety, Tolerability and Efficacy of MK-3475 in Combination With INCB024360 in Participants With Selected Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-202/ ECHO-202
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Microsatellite-instability (MSI) High Colorectal Cancer (CRC); Endometrial Cancer; Head and Neck Cancer; Hepatocellular Carcinoma (HCC); Gastric Cancer; Lung Cancer; Lymphoma; Renal Cell Carcinoma (RCC); Ovarian Cancer; Solid Tumors; UC (Urothelial Cancer); Melanoma; Bladder Cancer; Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Microsatellite Instability; Endometrial Neoplasms; Head and Neck Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Lung Neoplasms; Lymphoma; Carcinoma, Renal Cell; Ovarian Neoplasms; Melanoma; Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: MK-3475 + INCB024360 (Experimental): Phase 1: MK-3475 + INCB024360 25 mg twice a day (BID) as starting dose, followed by dose escalations (Phase 1) until recommended phase 2 dose of INCB024360 is determined
  Interventions: Drug: MK-3475; Drug: INCB024360
- Phase 2: MK-3475 + INCB024360 (Experimental): (recommended phase 2 dose)
  Interventions: Drug: MK-3475; Drug: INCB024360

INTERVENTIONS:
Drug: MK-3475 — IV infusion
Drug: INCB024360 — Oral daily dosing

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and efficacy when combining MK-3475 and INCB024360 in participants with certain cancers. This study was conducted in 2 phases, Phase 1 and Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically non-small cell lung cancer (NSCLC), melanoma, transitional cell carcinoma of the genitourinary (GU) tract, renal cell cancer, triple negative breast cancer, adenocarcinoma of the endometrium or squamous cell carcinoma of the head and neck (Phase 1).
* Subjects with histologically confirmed melanoma, NSCLC, transitional cell carcinoma of the GU tract, TNBC, SCCHN, ovarian cancer, MSI high colorectal cancer (CRC), RCC, gastric cancer, HCC and DLBCL (Phase 2).
* Life expectancy > 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Presence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Lugano Classification for subjects with DLBCL.
* Laboratory and medical history parameters within protocol-defined range.
* For Phase 1: Subjects who have advanced or metastatic disease as noted above that have received at least one prior therapy or have advanced or metastatic disease for which no curative treatment is available may be enrolled.
* For Phase 2 expansion cohorts: Subjects with NSCLC, melanoma (checkpoint inhibitor naïve, primary refractory melanoma, relapsed melanoma), transitional cell carcinoma of the GU tract, SCCHN, ovarian cancer, MSI high CRC, RCC, DLBCL, TNBC, gastric cancer, and HCC.

  * Phase 2 expansion: NSCLC

    * Subjects who have received at least 1 prior platinum-based therapy. Subjects who have a non-platinum-based regimen may be enrolled with medical monitor approval.
    * Tumors with epidermal growth factor receptor mutation positive or anaplastic lymphoma kinase fusion oncogene positive treated with a tyrosine kinase inhibitor are permitted; however, subjects should have progressed on or be intolerant to the targeted therapy.
    * Subjects must not have received immunotherapy with programmed death receptor-1 (PD-1) or cytotoxic T-lymphocyte antigen (CTLA-4) targeted therapy.
  * Phase 2 expansion: Melanoma

    * Documentation of V600E-activating BRAF mutation status.
    * Prior systemic therapy requirements.
    * Melanoma immune checkpoint-naïve: Subjects must not have received immunotherapy with anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy. Exception: Prior anti-CTLA-4 in the adjuvant setting would be permitted.
    * Primary refractory melanoma: Subjects must have received prior treatment with anti-PD-1 or anti-PD-L1 therapy (alone or as part of a combination) in the advanced or metastatic setting and have progressive disease as their best response to treatment that is confirmed 4 weeks later.
    * Relapsed melanoma: Subjects must have received prior anti-PD-1 or anti-PD-L1 therapy (alone or as part of a combination) in the advanced or metastatic setting and achieved partial response ore complete response but later have confirmed progressive disease.
    * Subjects enrolling in the primary refractory or relapsed melanoma must be willing to undergo mandatory pretreatment and on-treatment biopsies.
    * Ocular melanoma is excluded.
  * Phase 2 expansion: Transitional cell carcinoma of the GU tract

    * Metastatic or locally advanced and not amenable to curative therapy with disease progression on or after platinum-based chemotherapy or alternative therapy if platinum-based therapy is not appropriate.
    * Prior PD-1 or CTLA-4 targeted therapies are excluded
  * Phase 2 expansion: SCCHN

    * Histologically confirmed metastatic or recurrent squamous cell carcinoma not amenable to local therapy with curative intent (surgery or radiation with or without chemotherapy). Carcinoma of the nasopharynx, salivary gland, or * *Subjects must have received at least 1 prior systemic chemotherapy regimen that must have included a platinum-based therapy.
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
  * Phase 2 expansion: Ovarian cancer

    * Subjects with FIGO Stage Ic, Stage II, Stage III, Stage IV, recurrent, or persistent (unresectable) histologically confirmed epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube carcinoma.
    * Subjects must have received a platinum-taxane-based regimen as first-line therapy.
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
    * Borderline, low-malignant-potential epithelial carcinoma per histopathology is excluded.
  * Phase 2 expansion: Relapsed or refractory DLBCL

    * Prior allogeneic stem-cell transplantation is excluded.
    * Must have received > or = 1 prior treatment regimen.
    * Not a candidate for curative therapy or hematopoietic stem-cell transplantation (either due to disease burden, fitness, or preference).
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
  * Phase 2 expansion: TNBC

    * Histologically confirmed breast adenocarcinoma that is unresectable loco regional, or metastatic
    * Pathologically confirmed as triple negative, source documented, defined as both of the following:
    * Estrogen receptor (ER) and progesterone receptor (PgR) negative.
    * Human epidermal growth factor receptor 2 (HER2) negative as per American Society of Clinical Oncology/College of American Pathologists guidelines.
    * Subject must have received at least 1 prior systemic regimen for advanced or metastatic disease
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
  * Phase 2 expansion: RCC

    * Subjects with histological or cytological confirmation of clear cell RCC.
    * Not curable by surgery.
    * Subjects must have received prior antiangiogenic therapy.
    * Subjects must not have received prior immunotherapy with anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy.
  * Phase 2 expansion: MSI high CRC

    * Subjects with histological confirmation of locally advanced unresectable or metastatic MSI high CRC.
    * MSI status is, respectively, determined by examining CRC tumor.
    * Subjects may have received no more than 2 lines of prior therapy for advanced disease.
  * Phase 2 expansion: Gastric Cancer

    * Must have histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma.
    * Must have progression on or after therapy containing platinum/fluoropyrimidine or refused standard therapy.
    * Subjects may have received no more than 2 lines of prior therapy for advanced disease.
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
  * Phase 2 expansion: HCC

    * Must have histologically or cytologically confirmed diagnosis of HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible).
    * Barcelona Clinic Liver Cancer (BCLC) Stage C disease (Llovet et al 1999), or BCLC Stage B disease.
    * Subjects may have received no more than 2 lines of prior therapy for the advanced disease
    * Must have progressed on, refused, or were intolerant of sorafenib.
    * The following are excluded: Subjects with liver transplants, clear invasion of the bile duct or main portal branch(es), or hepatorenal syndrome, or subjects who have required esophageal variceal ablation within 28 days of starting study treatment.
    * Prior PD-1 or CTLA-4 targeted therapies are excluded.
  * Tumor biopsies are required. If a subject has inaccessible lesions, such as in ovarian cancer, HCC, or gastric cancer, or highly vascular lesions, such as RCC, enrollment may be considered with medical monitor approval, and archived tissue may be acceptable.
  * Females of child-bearing potential and males who use adequate birth control through 120 days post dose.

Exclusion Criteria:

* Subjects who participated in any other study in which receipt of an investigational study drug or device occurred within 2 weeks or 5 half-lives (whichever is longer) prior to first dose.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). Exception: Prior anti-CTLA-4 in the adjuvant setting for subjects with melanoma would be permitted.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable.
* Has an active autoimmune disease.
* Has evidence of noninfectious pneumonitis that required steroids or current pneumonitis.
* Live vaccine use within 30 days of first dose of study medication.
* Monoamine oxidase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (24):
- United States (24):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - US Davis Cancer Center, Sacramento, California
  - University Of Colorado Cancer Center, Aurora, Colorado
  - University of Connecticut Health Center Carole And Ray Neag Comprehensive Cancer Center, Farmington, Connecticut
  - Miami Cancer Institute at Baptist Health, Inc, Miami, Florida
  - Georgia Cancer Specialists affiliated with Northside Hospital Cancer Institute, Atlanta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - St. Francis Cancer Center, Topeka, Kansas
  - Greater Baltimore Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Institute, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders (RCCA MD LLC- Maryland Division), Bethesda, Maryland
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Health Partners Institute, Saint Louis Park, Minnesota
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - The Christ Hospital Hematology Oncology, Lindner Research Center, Cincinnati, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center At Dallas, Dallas, Texas
  - Virginia Cancer Specialists, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 22 investigative sites in the United States from 17July 2014 to 06 November 2020.
Pre-assignment Details: Prior to 17May18 study amended/discontinued, 444 participants were enrolled. Survival follow up and monotherapy option after discontinuation of combination were removed so anyone in survival follow up were discontinued the study and were assigned to "study terminated by sponsor" because completed was not an option in the database for those in survival follow up. 1 patient on combo treatment did not move to the monotherapy so they were also assigned to this reason for discontinuing.
Groups:
- Phase 1: Epacadostat 25 mg BID: Epacadostat 25 mg tablet orally twice daily (BID) starting on Cycle 1 Day 1 in combination with pembrolizumab 2 mg/kg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1.
- Phase 1: Epacadostat 50 mg BID: Epacadostat 50 mg tablet orally BID starting on Cycle 1 Day 1 in combination with pembrolizumab 2 mg/kg or 200mg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1.
- Phase 1: Epacadostat 100 mg BID: Epacadostat 100 mg tablet orally BID starting on Cycle 1 Day 1 in combination with pembrolizumab 2 mg/kg or 200mg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1.
- Phase 1: Epacadostat 300 mg BID: Epacadostat 300 mg tablet orally BID starting on Cycle 1 Day 1 in combination with pembrolizumab 200 mg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1.
- Phase 2: Epacadostat 100 mg BID: Epacadostat 100 mg tablet orally BID in combination with pembrolizumab 200 mg intravenously every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Phase 1: Epacadostat 25 mg BID | Phase 1: Epacadostat 50 mg BID | Phase 1: Epacadostat 100 mg BID | Phase 1: Epacadostat 300 mg BID | Phase 2: Epacadostat 100 mg BID
Started | 4 | 20 | 18 | 20 | 382
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 20 | 18 | 20 | 382
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 33
Not completed — Death | 2 | 13 | 12 | 12 | 205
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 11
Not completed — Study terminated by Sponsor | 2 | 7 | 6 | 4 | 128
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety evaluable population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Epacadostat 25 mg BID | Phase 1: Epacadostat 50 mg BID | Phase 1: Epacadostat 100 mg BID | Phase 1: Epacadostat 300 mg BID | Phase 2: Epacadostat 100 mg BID | Total
Number analyzed (Participants) | 4 | 20 | 18 | 20 | 382 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (18.01) | 60.8 (12.97) | 63.2 (13.67) | 59.2 (13.06) | 62.7 (11.60) | 62.3 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 6 | 9 | 181 | 208
  Male | 1 | 11 | 12 | 11 | 201 | 236
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 1 | 20 | 18 | 17 | 337 | 393
  Black/African-American | 1 | 0 | 0 | 2 | 19 | 22
  Asian | 1 | 0 | 0 | 1 | 15 | 17
  Native Hawaiian/Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 9 | 9
  Missing | 0 | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 16 | 18
  Not Hispanic or Latino | 4 | 20 | 17 | 19 | 353 | 413
  Unknown | 0 | 0 | 0 | 0 | 10 | 10
  Other | 0 | 0 | 0 | 0 | 2 | 2
  Missing | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE) and Serious Treatment-Emergent Adverse Events
Description: An adverse event is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after a participant provides informed consent. A TEAE is any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug. Serious adverse event (SAE) is defined as an event that meets 1 of the following criteria: is fatal or life threatening, results in persistent or significant disability or incapacity, constitutes a congenital anomaly or birth defect, is clinically meaningful (i.e. defined as an event that jeopardizes the participant or requires potential medical or surgical intervention to prevent 1 of the outcomes listed above) or requires inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: Approximately 54 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 1: Epacadostat 25 mg BID | Phase 1: Epacadostat 50 mg BID | Phase 1: Epacadostat 100 mg BID | Phase 1: Epacadostat 300 mg BID
Number analyzed (Participants) | 4 | 20 | 18 | 20
Percentage of Participants
  SAE | 0 | 40.0 | 50.0 | 45.0
  TEAS | 100. | 95.0 | 94.4 | 100.

2. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was percentage of participants with best overall response [complete response (CR) or partial response (PR)], per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Approximately 54 months
Population: The efficacy evaluable population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab). Number analyzed indicated participants analyzed in the respective tumor type.
Measure: Number; unit: percentage of participants
Groups:
- Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W: Epacadostat 100 mg tablet orally BID in combination with pembrolizumab 200 mg intravenously every 3 weeks (Q3W).
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 382
percentage of participants
  Triple negative breast cancer: number analyzed (Participants) | 36
  Triple negative breast cancer | 11.1
  Microsatellite-instability high colorectal cancer: number analyzed (Participants) | 16
  Microsatellite-instability high colorectal cancer | 43.8
  Gastric cancer: number analyzed (Participants) | 27
  Gastric cancer | 22.2
  Hepatocellular carcinoma: number analyzed (Participants) | 24
  Hepatocellular carcinoma | 16.7
  Melanoma - immune checkpoint-naïve: number analyzed (Participants) | 43
  Melanoma - immune checkpoint-naïve | 60.5
  Non-small cell lung cancer (NSCLC) (tumor proportion score (TPS) < 50% or indeterminate): number analyzed (Participants) | 13
  Non-small cell lung cancer (NSCLC) (tumor proportion score (TPS) < 50% or indeterminate) | 30.8
  NSCLC programmed cell death ligand (PD-L1) low negative (TPS < 50%): number analyzed (Participants) | 45
  NSCLC programmed cell death ligand (PD-L1) low negative (TPS < 50%) | 24.4
  Ovarian cancer: number analyzed (Participants) | 37
  Ovarian cancer | 8.1
  Renal cell carcinoma: number analyzed (Participants) | 37
  Renal cell carcinoma | 32.4
  Squamous cell carcinoma of the head and neck: number analyzed (Participants) | 36
  Squamous cell carcinoma of the head and neck | 33.3
  Transitional carcinoma of the genitourinary (GU) tract: number analyzed (Participants) | 36
  Transitional carcinoma of the genitourinary (GU) tract | 30.6
  Diffuse large B-cell lymphoma: number analyzed (Participants) | 26
  Diffuse large B-cell lymphoma | 19.2
  Primary Refractory Melanoma: number analyzed (Participants) | 3
  Primary Refractory Melanoma | 0.0
  Relapsed Melanoma: number analyzed (Participants) | 3
  Relapsed Melanoma | 0.0

3. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: Duration of response is the time from the first overall response contributing to an objective response (complete or partial response) for DLBCL to the date of death or the date of first overall response of progressive diseasemeasured (by irRECIST for solid tumors or the Lugano Classification, whichever is earliest.
Time Frame: Up to 54 months
Population: The efficacy evaluable population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab).
  Number analyzed indicated participants analyzed in the respective tumor type and those who responded.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W: Epacadostat 100 mg tablet orally BID starting on Cycle 1 Day 1 in combination with pembrolizumab 200 mg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1.
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 105
Months
  Hepatocellular Carcinoma: number analyzed (Participants) | 4
  Hepatocellular Carcinoma | NA [2.04 to NA] — insufficient number of participants with events
  Triple Negative Breast Cancer: number analyzed (Participants) | 4
  Triple Negative Breast Cancer | NA [0.92 to NA] — insufficient number of participants with events
  Immune Checkpoint-naïve Melanoma: number analyzed (Participants) | 26
  Immune Checkpoint-naïve Melanoma | NA [26.35 to NA] — insufficient number of participants with events
  NSCLC high positive (PD-L1 TPS ≥ 50%): number analyzed (Participants) | 4
  NSCLC high positive (PD-L1 TPS ≥ 50%) | 12.44 [2.10 to 16.53]
  NSCLC low/negative or indeterminate (PD-L1 TPS < 50% or indeterminate): number analyzed (Participants) | 2
  NSCLC low/negative or indeterminate (PD-L1 TPS < 50% or indeterminate) | 11.93 [8.90 to 14.95]
  NSCLC (TPS 0%): number analyzed (Participants) | 4
  NSCLC (TPS 0%) | NA [7.43 to NA] — insufficient number of participants with events
  NSCLC Unknown: number analyzed (Participants) | 5
  NSCLC Unknown | 10.84 [4.14 to NA] — insufficient number of participants with events
  Renal Cell Carcinoma: number analyzed (Participants) | 12
  Renal Cell Carcinoma | 16.95 [12.58 to NA] — insufficient number of participants with events
  Squamous Cell Carcinoma of the Head and Neck: number analyzed (Participants) | 12
  Squamous Cell Carcinoma of the Head and Neck | 11.33 [3.94 to 31.74]
  Transitional Cell Carcinoma of the GU Tract: number analyzed (Participants) | 11
  Transitional Cell Carcinoma of the GU Tract | NA [10.64 to NA] — insufficient number of participants with events
  Ovarian Cancer: number analyzed (Participants) | 3
  Ovarian Cancer | NA [5.75 to NA] — insufficient number of participants with events
  Gastric Cancer: number analyzed (Participants) | 6
  Gastric Cancer | NA [0.46 to NA] — insufficient number of participants with events
  MSI high Colorectal Cancer: number analyzed (Participants) | 7
  MSI high Colorectal Cancer | NA [4.17 to NA] — insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 5
  DLBCL | 3.66 [0.72 to NA] — insufficient number of participants with events

4. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: Progression-free survival is defined as number of days from the first day of taking study drug to the earlier of death or disease progression by irRECIST v1.1 for select solid tumors and modified Lugano Classification for DLBCL.
Time Frame: Up to 54 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 382
Months
  Hepatocellular Carcinoma: number analyzed (Participants) | 24
  Hepatocellular Carcinoma | 5.49 [2.69 to 10.28]
  Triple Negative Breast Cancer: number analyzed (Participants) | 36
  Triple Negative Breast Cancer | 1.97 [1.87 to 2.92]
  Immune Checkpoint-naïve Melanoma: number analyzed (Participants) | 43
  Immune Checkpoint-naïve Melanoma | 16.69 [6.24 to NA] — insufficient number of participants with events
  Primary Refractory Melanoma: number analyzed (Participants) | 3
  Primary Refractory Melanoma | 1.69 [1.25 to 2.14]
  Relapsed Melanoma: number analyzed (Participants) | 3
  Relapsed Melanoma | 2.60 [2.14 to 4.21]
  NSCLC: number analyzed (Participants) | 58
  NSCLC | 4.09 [2.14 to 7.36]
  Renal Cell Carcinoma: number analyzed (Participants) | 37
  Renal Cell Carcinoma | 4.50 [2.33 to 6.24]
  Squamous Cell Carcinoma of the Head and Neck: number analyzed (Participants) | 36
  Squamous Cell Carcinoma of the Head and Neck | 4.37 [2.30 to 7.79]
  Transitional Cell Carcinoma of the GU Tract: number analyzed (Participants) | 36
  Transitional Cell Carcinoma of the GU Tract | 4.40 [2.14 to 8.90]
  Ovarian Cancer: number analyzed (Participants) | 37
  Ovarian Cancer | 2.10 [1.97 to 2.83]
  Gastric Cancer: number analyzed (Participants) | 27
  Gastric Cancer | 1.97 [1.41 to 2.07]
  MSI high Colorectal Cancer: number analyzed (Participants) | 16
  MSI high Colorectal Cancer | 6.11 [2.07 to NA] — insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 26
  DLBCL | 2.63 [1.87 to 4.01]

5. Secondary Outcome: Phase 2: Duration of Disease Control
Description: The duration of disease control is the time from the treatment start date to the first objective response of PD (by irRECIST v1.1 or Lugano Classification), death, or last tumor assessment date (if PD/death not present), for subjects with best overall response of SD or better.
Time Frame: Up to 54 months
Population: The Efficacy Evaluable Population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab). Number analyzed indicated participants analyzed in the respective tumor type. The median time and the 90% CI were estimated using Kaplan-Meier method.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 191
Months
  Hepatocellular Carcinoma: number analyzed (Participants) | 15
  Hepatocellular Carcinoma | 10.38 [5.49 to NA] — insufficient number of participants with events
  Triple Negative Breast Cancer: number analyzed (Participants) | 11
  Triple Negative Breast Cancer | 11.47 [4.01 to 12.65]
  Immune Checkpoint-naïve Melanoma: number analyzed (Participants) | 31
  Immune Checkpoint-naïve Melanoma | 30.29 [25.03 to NA] — insufficient number of participants with events
  Relapsed Melanoma: number analyzed (Participants) | 1
  Relapsed Melanoma | 4.21 [NA to NA] — insufficient number of participants with events
  NSCLC Total: number analyzed (Participants) | 30
  NSCLC Total | 14.42 [8.51 to 19.45]
  Renal Cell Carcinoma: number analyzed (Participants) | 22
  Renal Cell Carcinoma | 13.39 [5.13 to 18.86]
  Squamous Cell Carcinoma of the Head and Neck: number analyzed (Participants) | 20
  Squamous Cell Carcinoma of the Head and Neck | 9.18 [6.24 to 13.34]
  Transitional Cell Carcinoma of the GU Tract: number analyzed (Participants) | 21
  Transitional Cell Carcinoma of the GU Tract | 15.36 [8.41 to 22.74]
  Ovarian Cancer: number analyzed (Participants) | 14
  Ovarian Cancer | 5.08 [3.29 to 7.79]
  Gastric Cancer: number analyzed (Participants) | 7
  Gastric Cancer | NA [2.56 to NA] — insufficient number of participants with events
  MSI high Colorectal Cancer: number analyzed (Participants) | 10
  MSI high Colorectal Cancer | NA [6.11 to NA] — insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 9
  DLBCL | 7.29 [4.01 to 10.91]

6. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival is determined from the date of first dose until death due to any cause.
Time Frame: Up to 54 months
Population: The Efficacy Evaluable Population included all participants enrolled in the study who received at least 1 dose of study drug. Number analyzed indicated participants analyzed in the respective tumor type. The median time and the 90% CI were estimated using Kaplan-Meier method.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 382
Months
  Hepatocellular Carcinoma: number analyzed (Participants) | 24
  Hepatocellular Carcinoma | NA [8.94 to NA] — insufficient number of participants with events
  Triple Negative Breast Cancer: number analyzed (Participants) | 36
  Triple Negative Breast Cancer | 5.16 [4.60 to 7.46]
  Immune Checkpoint-naïve Melanoma: number analyzed (Participants) | 43
  Immune Checkpoint-naïve Melanoma | NA [NA to NA] — insufficient number of participants with events
  Primary Refractory Melanoma: number analyzed (Participants) | 3
  Primary Refractory Melanoma | NA [NA to NA] — insufficient number of participants with events
  Relapsed Melanoma: number analyzed (Participants) | 3
  Relapsed Melanoma | NA [2.60 to NA] — insufficient number of participants with events
  NSCLC: number analyzed (Participants) | 58
  NSCLC | 14.62 [9.72 to 24.38]
  Renal Cell Carcinoma: number analyzed (Participants) | 37
  Renal Cell Carcinoma | NA [18.40 to NA] — insufficient number of participants with events
  Squamous Cell Carcinoma of the Head and Neck: number analyzed (Participants) | 36
  Squamous Cell Carcinoma of the Head and Neck | 8.34 [4.37 to 15.41]
  Transitional Cell Carcinoma of the GU Tract: number analyzed (Participants) | 36
  Transitional Cell Carcinoma of the GU Tract | 13.44 [8.41 to NA] — insufficient number of participants with events
  Ovarian Cancer: number analyzed (Participants) | 37
  Ovarian Cancer | 13.11 [8.34 to 25.92]
  Gastric Cancer: number analyzed (Participants) | 27
  Gastric Cancer | 4.04 [1.97 to 15.84]
  MSI high Colorectal Cancer: number analyzed (Participants) | 16
  MSI high Colorectal Cancer | NA [8.15 to NA] — insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 26
  DLBCL | 11.79 [4.37 to NA] — insufficient number of participants with events

7. Secondary Outcome: Phase 2: Ordinal Categorical Response Score
Description: Ordinal categorical response score, determined by radiographic disease assessments per irRECIST v1.1. The 5-category ordinal response endpoint is determined at a given timepoint by classifying response into one of the following groups: 1 = Complete response per irRECIST v1.1 2 = Very good response, defined as > 60% tumor reduction 3 = Minor response, defined as > 30% to ≤ 60% tumor reduction 4 = Stable disease per irRECIST v1.1 5 = Progressive disease per irRECIST v1.1
Time Frame: Up to 54 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Epacadostat 100 mg BID+ Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 382
Participants
  Hepatocellular Carcinoma: number analyzed (Participants) | 24
  Hepatocellular Carcinoma: Complete Response - Score 1 | 0
  Hepatocellular Carcinoma: Very Good Response - Score 2 | 2
  Hepatocellular Carcinoma: Minor Response - Score 3 | 2
  Hepatocellular Carcinoma: Stable Disease - Score 4 | 11
  Hepatocellular Carcinoma: Progressive Disease - Score 5 | 8
  Hepatocellular Carcinoma: Unable to Evaluable | 1
  Triple Negative Breast Cancer: number analyzed (Participants) | 36
  Triple Negative Breast Cancer: Complete Response - Score 1 | 1
  Triple Negative Breast Cancer: Very Good Response - Score 2 | 1
  Triple Negative Breast Cancer: Minor Response - Score 3 | 2
  Triple Negative Breast Cancer: Stable Disease - Score 4 | 7
  Triple Negative Breast Cancer: Progressive Disease - Score 5 | 19
  Triple Negative Breast Cancer: Unable to Evaluable | 6
  Immune Checkpoint-naïve Melanoma: number analyzed (Participants) | 43
  Immune Checkpoint-naïve Melanoma: Complete Response - Score 1 | 3
  Immune Checkpoint-naïve Melanoma: Very Good Response - Score 2 | 17
  Immune Checkpoint-naïve Melanoma: Minor Response - Score 3 | 6
  Immune Checkpoint-naïve Melanoma: Stable Disease - Score 4 | 5
  Immune Checkpoint-naïve Melanoma: Progressive Disease - Score 5 | 10
  Immune Checkpoint-naïve Melanoma: Unable to Evaluable | 2
  Primary Refractory Melanoma: number analyzed (Participants) | 3
  Primary Refractory Melanoma: Complete Response - Score 1 | 0
  Primary Refractory Melanoma: Very Good Response - Score 2 | 0
  Primary Refractory Melanoma: Minor Response - Score 3 | 0
  Primary Refractory Melanoma: Stable Disease - Score 4 | 0
  Primary Refractory Melanoma: Progressive Disease - Score 5 | 2
  Primary Refractory Melanoma: Unable to Evaluable | 1
  Relapsed Melanoma: number analyzed (Participants) | 36
  Relapsed Melanoma: Complete Response - Score 1 | 3
  Relapsed Melanoma: Very Good Response - Score 2 | 4
  Relapsed Melanoma: Minor Response - Score 3 | 5
  Relapsed Melanoma: Stable Disease - Score 4 | 8
  Relapsed Melanoma: Progressive Disease - Score 5 | 10
  Relapsed Melanoma: Unable to Evaluable | 6
  NSCLC: number analyzed (Participants) | 58
  NSCLC: Complete Response - Score 1 | 4
  NSCLC: Very Good Response - Score 2 | 3
  NSCLC: Minor Response - Score 3 | 8
  NSCLC: Stable Disease - Score 4 | 15
  NSCLC: Progressive Disease - Score 5 | 24
  NSCLC: Unable to Evaluable | 4
  Renal Cell Carcinoma: number analyzed (Participants) | 37
  Renal Cell Carcinoma: Complete Response - Score 1 | 2
  Renal Cell Carcinoma: Very Good Response - Score 2 | 6
  Renal Cell Carcinoma: Minor Response - Score 3 | 4
  Renal Cell Carcinoma: Stable Disease - Score 4 | 10
  Renal Cell Carcinoma: Progressive Disease - Score 5 | 13
  Renal Cell Carcinoma: Unable to Evaluable | 2
  Squamous Cell Carcinoma of the Head and Neck: number analyzed (Participants) | 36
  Squamous Cell Carcinoma of the Head and Neck: Complete Response - Score 1 | 3
  Squamous Cell Carcinoma of the Head and Neck: Very Good Response - Score 2 | 4
  Squamous Cell Carcinoma of the Head and Neck: Minor Response - Score 3 | 5
  Squamous Cell Carcinoma of the Head and Neck: Stable Disease - Score 4 | 8
  Squamous Cell Carcinoma of the Head and Neck: Progressive Disease - Score 5 | 10
  Squamous Cell Carcinoma of the Head and Neck: Unable to Evaluable | 6
  Transitional Cell Carcinoma of the GU Tract: number analyzed (Participants) | 36
  Transitional Cell Carcinoma of the GU Tract: Complete Response - Score 1 | 2
  Transitional Cell Carcinoma of the GU Tract: Very Good Response - Score 2 | 4
  Transitional Cell Carcinoma of the GU Tract: Minor Response - Score 3 | 5
  Transitional Cell Carcinoma of the GU Tract: Stable Disease - Score 4 | 10
  Transitional Cell Carcinoma of the GU Tract: Progressive Disease - Score 5 | 11
  Transitional Cell Carcinoma of the GU Tract: Unable to Evaluable | 4
  Ovarian Cancer: number analyzed (Participants) | 37
  Ovarian Cancer: Complete Response - Score 1 | 1
  Ovarian Cancer: Very Good Response - Score 2 | 0
  Ovarian Cancer: Minor Response - Score 3 | 2
  Ovarian Cancer: Stable Disease - Score 4 | 11
  Ovarian Cancer: Progressive Disease - Score 5 | 16
  Ovarian Cancer: Unable to Evaluable | 7
  Gastric Cancer: number analyzed (Participants) | 27
  Gastric Cancer: Complete Response - Score 1 | 0
  Gastric Cancer: Very Good Response - Score 2 | 1
  Gastric Cancer: Minor Response - Score 3 | 5
  Gastric Cancer: Stable Disease - Score 4 | 1
  Gastric Cancer: Progressive Disease - Score 5 | 11
  Gastric Cancer: Unable to Evaluable | 9
  MSI high Colorectal Cancer: number analyzed (Participants) | 16
  MSI high Colorectal Cancer: Complete Response - Score 1 | 1
  MSI high Colorectal Cancer: Very Good Response - Score 2 | 3
  MSI high Colorectal Cancer: Minor Response - Score 3 | 3
  MSI high Colorectal Cancer: Stable Disease - Score 4 | 3
  MSI high Colorectal Cancer: Progressive Disease - Score 5 | 5
  MSI high Colorectal Cancer: Unable to Evaluable | 1

8. Secondary Outcome: Phase 2: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE) and Serious Treatment-Emergent Adverse Events
Time Frame: Up to 54 months
Population: The safety evaluable population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab). Treatment groups for this population were determined according to the actual treatment the participant receives on Day 1. All safety analyses were conducted using the safety evaluable population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Epacadostat 100 mg BID
Number analyzed (Participants) | 382
Percentage of Participants
  Treatment-Emergent Adverse Events (TEAE) | 100
  Serious Treatment-Emergent Adverse Events | 51.0

ADVERSE EVENTS:
Time Frame: Approximately 54 months
Description: The safety evaluable population included all participants enrolled in the study who received at least 1 dose of study drug (epacadostat or pembrolizumab).
Groups:
- Phase 1: Epacadostat 300 MG BID: Epacadostat 300 mg tablet orally BID starting on Cycle 1 Day 1 in combination with pembrolizumab 2 mg/kg or 200mg administered intravenously every 3 weeks (Q3W) starting on Cycle 1 Day 1
- Total: Total
Arm/Group | Phase 1: Epacadostat 25 mg BID | Phase 1: Epacadostat 50 MG BID | Phase 1: Epacadostat 100 MG BID | Phase 1: Epacadostat 300 MG BID | Phase 2: Epacadostat 100 MG BID | Total
All-Cause Mortality (participants affected / at risk) | 2/4 | 13/20 | 12/18 | 14/20 | 209/382 | 250/444
Serious Adverse Events (participants affected / at risk) | 0/4 | 8/20 | 9/18 | 9/20 | 195/382 | 221/444
Other Adverse Events (participants affected / at risk) | 4/4 | 18/20 | 17/18 | 20/20 | 375/382 | 434/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Epacadostat 25 mg BID (N=4) | Phase 1: Epacadostat 50 MG BID (N=20) | Phase 1: Epacadostat 100 MG BID (N=18) | Phase 1: Epacadostat 300 MG BID (N=20) | Phase 2: Epacadostat 100 MG BID (N=382) | Total (N=444)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 12 (13) | 14 (15)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 7 (8)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 5 (6)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (5)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 7 (7)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 6 (6)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 10 (10)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (9) | 11 (11)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 6 (7)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 33 (33) | 35 (35)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (13) | 13 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 11 (11) | 12 (12)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 15 (16) | 16 (17)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 7 (7)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 8 (8) | 10 (12)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 11 (12)
Spinal cord haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 10 (11)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Epacadostat 25 mg BID (N=4) | Phase 1: Epacadostat 50 MG BID (N=20) | Phase 1: Epacadostat 100 MG BID (N=18) | Phase 1: Epacadostat 300 MG BID (N=20) | Phase 2: Epacadostat 100 MG BID (N=382) | Total (N=444)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 12 (13)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 19 (19) | 25 (25)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 53 (60) | 59 (68)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 23 (25) | 25 (27)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (7) | 7 (9)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 36 (46) | 42 (54)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 9 (9)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 1 (5) | 2 (3) | 35 (45) | 39 (54)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 2 (6) | 3 (4) | 48 (65) | 55 (78)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 23 (24) | 31 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 9 (12) | 4 (6) | 6 (8) | 64 (88) | 87 (121)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 4 (6) | 1 (1) | 44 (56) | 51 (66)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (1) | 2 (3) | 1 (1) | 4 (4) | 27 (28) | 35 (37)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4) | 7 (8) | 5 (6) | 48 (58) | 65 (78)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 31 (37) | 36 (42)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 8 (8)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 25 (29) | 27 (32)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 6 (6)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (5) | 6 (7)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 11 (11)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 8 (8)
Cerebral cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Chest discomfort (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 10 (10)
Chills (General disorders) | 0 (0) | 4 (4) | 2 (3) | 3 (3) | 36 (40) | 45 (50)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 9 (9)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (4) | 8 (13) | 4 (4) | 3 (5) | 86 (94) | 104 (120)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (9) | 3 (3) | 9 (9) | 100 (114) | 122 (139)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 9 (9) | 95 (103) | 109 (117)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 32 (34) | 34 (36)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 18 (20) | 24 (26)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 5 (9) | 7 (12) | 5 (10) | 99 (142) | 119 (179)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 5 (9) | 2 (2) | 3 (4) | 40 (49) | 50 (64)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 24 (26) | 33 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 16 (18) | 20 (22)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 8 (8) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 12 (13)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (13) | 14 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 10 (11) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 6 (7) | 5 (7) | 69 (77) | 84 (96)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 20 (23) | 22 (25)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 8 (8)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 12 (13) | 15 (16)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 1 (3) | 2 (2) | 8 (9) | 13 (18)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 23 (24) | 26 (27)
Fatigue (General disorders) | 3 (5) | 13 (17) | 9 (10) | 13 (20) | 185 (220) | 223 (272)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 17 (19) | 21 (23)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 12 (14)
Foreign body reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (3) | 13 (13) | 19 (21)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (8) | 9 (10)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 7 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 11 (12) | 13 (14)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 6 (13) | 1 (1) | 4 (5) | 58 (77) | 71 (100)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 7 (7)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 9 (9)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 14 (14) | 16 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (4) | 3 (5) | 23 (31) | 29 (42)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 10 (11) | 12 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (3) | 21 (26) | 26 (34)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (5)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 9 (9) | 11 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 15 (17) | 16 (18)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 12 (13) | 17 (19)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 14 (14) | 17 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 11 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 6 (6) | 8 (9)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 30 (39) | 34 (43)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 12 (17) | 14 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 39 (57) | 43 (63)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 17 (25) | 19 (31)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 11 (14) | 12 (15)
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 29 (30) | 32 (33)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Influenza (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 9 (11) | 11 (15)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 15 (15) | 17 (17)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 6 (6) | 1 (1) | 2 (2) | 44 (48) | 55 (59)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 3 (13) | 3 (6) | 48 (80) | 54 (99)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 8 (9)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 7 (8)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 23 (31) | 25 (33)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 16 (16) | 19 (19)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 13 (16) | 15 (18)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 28 (30) | 36 (39)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 4 (4) | 10 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3) | 5 (7) | 22 (25) | 34 (39)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 20 (22) | 25 (27)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (12) | 0 (0) | 1 (1) | 24 (24) | 30 (38)
Nausea (Gastrointestinal disorders) | 3 (6) | 9 (20) | 5 (5) | 11 (18) | 115 (143) | 143 (192)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 12 (12) | 14 (14)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 14 (14) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 5 (7)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 31 (32) | 34 (35)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 7 (7)
Oedema peripheral (General disorders) | 1 (1) | 3 (4) | 3 (5) | 2 (2) | 40 (46) | 49 (58)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 19 (21) | 24 (28)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 17 (19) | 21 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 0 (0) | 5 (7) | 40 (45) | 51 (60)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (10) | 11 (12)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 8 (9)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (8) | 10 (10)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 9 (11) | 10 (13)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 10 (11) | 12 (13)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 6 (7)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 14 (16) | 17 (19)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 9 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 25 (28) | 31 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (12) | 2 (2) | 9 (12) | 78 (96) | 98 (126)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 6 (6)
Pyrexia (General disorders) | 0 (0) | 3 (5) | 3 (4) | 9 (10) | 58 (74) | 73 (93)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (10) | 1 (1) | 6 (13) | 86 (108) | 101 (135)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 4 (5) | 19 (23) | 26 (32)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (11) | 11 (11) | 15 (24)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 8 (8) | 11 (12)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 9 (9)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 10 (10) | 13 (13)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 6 (7)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 21 (25) | 23 (27)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 8 (10) | 12 (14)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Slow speech (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (3) | 11 (13) | 15 (20)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 11 (13) | 16 (19)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 10 (10) | 12 (12)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 5 (6)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (6)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 7 (7)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (6) | 2 (2) | 2 (2) | 31 (38) | 38 (48)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 10 (10) | 14 (14)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (8) | 0 (0) | 1 (1) | 28 (36) | 32 (47)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 14 (14) | 16 (16)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (5) | 4 (8) | 10 (13) | 78 (99) | 97 (127)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 35 (37) | 40 (42)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 8 (9) | 10 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 16 (18) | 19 (21)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 14 (16) | 15 (17)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Study enrollment was permanently discontinued on 17 May 2018 as a strategic decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT02178722/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT02178722/SAP_001.pdf